CLINICAL TRIAL: NCT04424966
Title: A Phase 0 Study of Infigratinib in Recurrent High-Grade Glioma Participants Scheduled for Resection to Evaluate Central Nervous System (CNS) Penetration With PK Triggered Expansion Cohort
Brief Title: Infigratinib in Recurrent High-Grade Glioma Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study drug no longer available.
Sponsor: Nader Sanai (Other)
Collaborators: Ivy Brain Tumor Center (Other); Barrow Neurological Institute (Other); QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor-Investigator, Nader Sanai, Deputy Director, Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-08; 20-500-092-34-38 (Other: SJHMC)
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Glioma; Glioblastoma; GBM
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Phase 0: 125 mg of infigratinib administered orally for 7 days prior to surgical resection.
  Expansion Cohort: 125 mg of infigratinib administered orally for 21 days of a 28-day treatment cycles.
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — The Phase 0 study will include treatment of recurrent high-grade glioma participants with 125 mg of infigratinib 7 days prior to surgical resection. Participants with tumors demonstrating PK-response will continue treatment with the same dose continuously for 21 days in 28-day cycles after surgery.

SUMMARY:
This trial is an open-label, multicenter, Phase 0 trial that will enroll up to 20 participants with recurrent high-grade glioma with FGFR1 K656E or FGFR3 K650E mutation or FGFR3-TACC3 translocation which are scheduled for resection. In the lead-in cohort, a total of 20 participants will be enrolled into the proposed phase 0 clinical trial. Participants will be administered infigratinib prior to surgical resection of their tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Prior resection of histologically diagnosed high-grade gliomas (III and IV) defined as participants who have progressed on or following standard (Stupp regimen) therapy, which included maximal surgical resection, temozolomide, and fractionated radiotherapy.
2. Recurrence must be confirmed by diagnostic biopsy with local pathology review or contrast-enhanced MRI.
3. Have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm, as per RANO criteria.
4. Sufficient archival tissue available to confirm eligibility.
5. Archival tissue must demonstrate: FGFR1 K656E or FGFR3 K650E mutation or FGFR3-TACC3 translocation from NGS sequencing or IHC and RT-PCR.
6. Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
7. Has voluntarily agreed to participate by giving written informed consent (personally or via legally authorized representative(s), and assent if applicable). Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
8. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
9. Age ≥18 at time of consent
10. Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology (Group (ECOG) scale (Oken et al. 1982)
11. Ability to swallow oral medications.
12. Has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

    1. Adequate bone marrow function:

       * absolute neutrophil count ≥1,000/mcL
       * Platelets (at time of surgery) ≥100,000/mcL
       * hemoglobin ≥8.0 g/dL Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator.
    2. Adequate hepatic and renal function:

       * total bilirubin ≤1.5 X ULN Participants with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
       * AST(SGOT) ≤3 X institutional ULN
       * ALT(SGPT) ≤3 X institutional ULN
       * Calculated or measured creatinine clearance ≥45 mL/min
    3. Other Lab Values:

       * Amylase or lipase ≤2 X institutional ULN
       * calcium or phosphorus, or calcium-phosphorus product <55 mg2/dL2

    <!-- -->

    1. Inorganic phosphorus within normal limits
    2. Total corrected serum calcium within normal limits
13. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant has had a hysterectomy.
14. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 3 months after the end of treatment administration.
15. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and for an additional 1 month after the end of treatment administration. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner to prevent delivery of the drug via seminal fluid.
16. Agreement to adhere to Lifestyle Considerations throughout study duration.
17. Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to Day 1. A washout period of at least 21 days is required between last chemotherapy dose and Day 1 (provided the patient did not receive radiotherapy).
18. Participants who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and Day 1.

Exclusion Criteria:

1. Have a history of liver transplant.
2. Have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
3. Known active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
4. Have a history and/or current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium, vascular system, and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcification.
5. Have current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, inflammation or ulceration, keratoconjunctivitis confirmed by ophthalmic examination. Subjects with asymptomatic ophthalmic conditions assessed by the investigator to pose minimal risk for study participation may be enrolled in the study.
6. Have current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc.
7. Have had a recent (≤3 months prior to first dose of study drug) transient ischemic attack or stroke.
8. CTCAE (v5.0) Grade ≥2 hearing loss.
9. CTCAE (v5.0) Grade ≥2 neuropathy.
10. Have clinically significant cardiac disease including any of the following:

    1. Known congestive heart failure requiring treatment (New York Heart Association Grade ≥2), LVEF <50% or local lower limit of normal as determined by MUGA scan or echocardiogram (ECHO), or uncontrolled hypertension (refer to the European Society of Cardiology and European Society of Hypertension guidelines [Williams et al 2018]).
    2. Presence of Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≥2 ventricular arrhythmias, atrial fibrillation, bradycardia, or conduction abnormality.
    3. Unstable angina pectoris or acute myocardial infarction ≤3 months prior to first dose of study drug.
    4. QTcF >470 msec (males and females). Note: If the QTcF is >470 msec in the first ECG, a total of 3 ECGs separated by at least 5 minutes should be performed. If the average of these 3 consecutive results for QTcF is ≤470 msec, the participant meets eligibility in this regard.
    5. Known history of congenital long QT syndrome.
11. Has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
12. Prior therapy with any mitogen-activated protein kinase (MEK) or FGFR inhibitor. Prior therapy is defined as a therapeutic dosing, as determined by the Investigator.
13. Are currently receiving or are planning to receive during participation in this study, treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration. Participants are not permitted to receive enzyme-inducing anti-epileptic drugs, including carbamazepine, phenytoin, phenobarbital, and primidone.
14. Current use of coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
15. Have any known hypersensitivity to gemcitabine, cisplatin, calcium-lowering agents, infigratinib, or their excipients.
16. Treatment with another investigational drug or other intervention within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
17. Have consumed grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges or products containing juice of these fruits within 7 days prior to first dose of study drug.
18. Have used medications known to prolong the QT interval and/or are associated with a risk of Torsades de Pointes (TdP) 7 days prior to first dose of study drug.
19. Have used amiodarone within 90 days prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ivy Brain Tumor Center Website — https://www.ivybraintumorcenter.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Recurrent High Grade Glioma: Participants with recurrent high grade glioma with FGFR1 K656E mutation, or FGFR3 K650E mutation, or FGFR3-TACC3 translocation who are scheduled for surgical resection.
  125 mg of infigratinib will be administered orally for 7 days prior to surgical resection during the Phase 0 component. Participants with tumors demonstrating positive PK response will continue treatment in the expansion phase component.
  125 mg of infigratinib will be administered orally for 21 consecutive days during 28-day treatment cycles during the expansion phase component.
Period: Phase 0
Arm/Group | Recurrent High Grade Glioma
Started | 7
Completed | 7
Not Completed | 0
Period: Expansion Phase
Arm/Group | Recurrent High Grade Glioma
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recurrent High Grade Glioma
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 63 [48 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Concentration of Infigratinib in Enhancing and Non-Enhancing Tumor Tissue
Description: Phase 0: Total infigratinib concentration in Gd enhancing and Gd non-enhancing tumor tissue collected intraoperatively, approximately 8 hours after study drug administration, will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Intraoperative
Measure: Geometric Mean (Full Range); unit: nM
Groups:
- Arm 1: Phase 0: 125 mg of infigratinib administered orally for 7 days prior to surgical resection.
  Expansion Cohort: 125 mg of infigratinib administered orally for 21 days of a 28-day treatment cycles.
  Infigratinib: The Phase 0 study will include treatment of recurrent high-grade glioma participants with 125 mg of infigratinib 7 days prior to surgical resection. Participants with tumors demonstrating PK-response will continue treatment with the same dose continuously for 21 days in 28-day cycles after surgery.
Arm/Group | Arm 1
Number analyzed (Participants) | 7
nM
  Total Concentration of Infigratinib in Enhancing Tissue | 790.6 [425.0 to 1259.1]
  Total Concentration of Infigratinib in Non-enhancing Tissue | 628.4 [86.4 to 1524.5]

2. Primary Outcome: Unbound Concentration of Infigratinib in Enhancing and Non-Enhancing Tumor Tissue
Description: Phase 0: Unbound infigratinib concentration in Gd enhancing and Gd non-enhancing tumor tissue collected intraoperatively, approximately 8 hours after study drug administration, will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Intraoperative
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Arm 1
Number analyzed (Participants) | 7
nM
  Unbound Concentration of Infigratinib in Enhancing Tissue | 4.4 [1.2 to 9.1]
  Unbound Concentration of Infigratinib in Non-enhancing Tissue | 3.5 [0.7 to 11.3]

3. Primary Outcome: Total Concentration of Infigratinib in Plasma
Description: Phase 0: Total infigratinib concentration in blood plasma collected intraoperatively, approximately 8 hours after study drug administration, will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Intraoperative
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Arm 1
Number analyzed (Participants) | 7
nM
  Total Concentration of Infigratinib in Plasma | 146.1 [56.4 to 334.3]
  Unbound Concentration of Infigratinib in Plasma | 0.8 [0.4 to 2.6]

4. Primary Outcome: Unbound Concentration of Infigratinib in Plasma
Description: Phase 0: Unbound infigratinib concentration in blood plasma collected intraoperatively, approximately 8 hours after study drug administration, will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Intraoperative
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Arm 1
Number analyzed (Participants) | 7
nM | 0.8 [0.4 to 2.6]

5. Primary Outcome: Total Concentration of Infigratinib in Cerebrospinal Fluid (CSF)
Description: Phase 0: Total infigratinib concentration in cerebrospinal fluid (CSF) collected intraoperatively, approximately 8 hours after study drug administration, will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Intraoperative
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Arm 1
Number analyzed (Participants) | 7
nM
  Total Concentration of Infigratinib in CSF | 7.1 [1.6 to 38.3]
  Unbound Concentration of Infigratinib in CSF | 7.1 [1.6 to 38.3]

6. Primary Outcome: Unbound Concentration of Infigratinib in Cerebrospinal Fluid (CSF)
Description: Phase 0: Unbound infigratinib concentration in cerebrospinal fluid (CSF) collected intraoperatively, approximately 8 hours after study drug administration, will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Intraoperative
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | Arm 1
Number analyzed (Participants) | 7
nM | 7.1 [1.6 to 38.3]

7. Primary Outcome: 6-month Progression-Free Survival (PFS6) in Expansion Phase Participants
Description: Proportion of participants who remain alive without disease progression at 6 months
Time Frame: From the date of Phase 0 surgery until the first documentation of disease progression or death due to any cause, assessed up to 6 months
Population: Participants who enrolled into the expansion phase component of the study. Participants alive without progression at 6 months were censored for PFS at the date of their last tumor assessment.
Measure: Number; unit: Percent
Arm/Group | Recurrent High Grade Glioma
Number analyzed (Participants) | 3
Percent | 66.7

8. Secondary Outcome: Mean % Change of pERK+ Cells in Resected Post-Treatment Recurrent HGG Tissue vs Baseline Tissue
Description: Phase 0: The mean percentage change of pERK positive cells in resected post-treatment recurrent high-grade glioma tumor tissue compared to baseline (archival primary high-grade glioma tumor tissue collected at screening) will be quantified using immunohistochemistry.
Time Frame: Baseline, Intraoperatively
Population: 1 participant was not assessed due to insufficient tissue for analysis.
Measure: Mean (Full Range); unit: Percentage of cells
Arm/Group | Recurrent High Grade Glioma
Number analyzed (Participants) | 6
Percentage of cells | 17.31 [-27.08 to 92.61]

9. Secondary Outcome: Mean % Change of MIB-1+ Cells in Resected Post-Treatment Recurrent HGG Tissue vs Baseline Tissue
Description: Phase 0: The mean percentage change of MIB-1 positive cells in resected post-treatment recurrent high-grade glioma tumor tissue compared to baseline (archival primary high-grade glioma tumor tissue collected at screening) will be quantified using immunohistochemistry.
Time Frame: Baseline, Intraoperatively
Population: 1 participant was not assessed due to insufficient tissue for analysis.
Measure: Mean (Full Range); unit: Percentage of cells
Arm/Group | Arm 1
Number analyzed (Participants) | 6
Percentage of cells | -7.39 [-17.28 to 2.88]

10. Secondary Outcome: Mean % Change of ClCas3+ Cells in Resected Post-Treatment Recurrent HGG Tissue vs Baseline Tissue
Description: Phase 0: The mean percentage change of ClCase3 positive cells in resected post-treatment recurrent high-grade glioma tumor tissue compared to baseline (archival primary high-grade glioma tumor tissue collected at screening) will be quantified using immunohistochemistry.
Time Frame: Baseline, Intraoperatively
Population: 1 participant was not assessed due to insufficient tissue for analysis.
Measure: Mean (Full Range); unit: Percentage of cells
Arm/Group | Arm 1
Number analyzed (Participants) | 6
Percentage of cells | 0.19 [-27.71 to 35.48]

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Assessed by CTCAE v5.0
Description: Expansion Phase: An AE that began after the start of study medication treatment; or if the event was continuous from baseline and was serious, study medication-related, or resulted in death, discontinuation, or interruption or reduction of trial therapy.
Time Frame: From date of first dose until 7 days after last dose, assessed over 2 years 6 months
Population: The analysis population includes participants who took at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent High Grade Glioma
Number analyzed (Participants) | 7
Participants | 5

12. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (TRAEs) Assessed by CTCAE v5.0
Description: Expansion Phase: TRAEs are those deemed definitely, probably, and potentially related to the study drug.
Time Frame: From date of first dose until 7 days after last dose, assessed over 2 years 6 months
Population: The analysis population includes participants who took at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent High Grade Glioma
Number analyzed (Participants) | 7
Participants | 5

13. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Expansion Phase: AE severity as defined according to CTCAE v5.0.
Time Frame: From date of first dose until 30 days after last dose, assessed over 2 years 6 months
Population: The analysis population includes participants who took at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent High Grade Glioma
Number analyzed (Participants) | 7
Participants | 0

14. Other Pre Specified Outcome: Total Infigratinib Peak Plasma Concentration (Cmax)
Description: Phase 0: Total infigratinib peak plasma concentration (Cmax) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Unbound Infigratinib Peak Plasma Concentration (Cmax)
Description: Phase 0: Unbound infigratinib peak plasma concentration (Cmax) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Total Infigratinib Time to Peak Plasma Concentration (Tmax)
Description: Phase 0: Total infigratinib time to peak plasma concentration (Tmax) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Unbound Infigratinib Time to Peak Plasma Concentration (Tmax)
Description: Phase 0: Unbound infigratinib time to peak plasma concentration (Tmax) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Total Infigratinib Concentration Half-Life (T1/2)
Description: Phase 0: Total infigratinib concentration half-life (T1/2) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Unbound Infigratinib Concentration Half-Life (T1/2)
Description: Phase 0: Unbound infigratinib concentration half-life (T1/2) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Total Infigratinib Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Phase 0: Total infigratinib area under the plasma concentration versus time curve (AUC) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Unbound Infigratinib Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Phase 0: Unbound infigratinib area under the plasma concentration versus time curve (AUC) in blood plasma will be determined by a validated liquid chromatography-mass spectrometry (LC-MS) method.
Time Frame: Day of surgery at pre-dose and 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Median Overall Survival (OS)
Description: Expansion Phase: The number of days from the date of Phase 0 surgery until the date of death due to any cause.
Time Frame: From the date of Phase 0 surgery until the date of death due to any cause, assessed over 2 years 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the day of first enrollment until 7 days after the final participant's final visit, approximately 2 years 6 months
Arm/Group | Recurrent High Grade Glioma
All-Cause Mortality (participants affected / at risk) | 6/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recurrent High Grade Glioma (N=7)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT04424966/Prot_SAP_000.pdf